CLINICAL TRIAL: NCT03584854
Title: Second-Line Uterotonics in Postpartum Hemorrhage: A Randomized Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jimin Kim, MD, Attending anesthesiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018P000775-A
Record Dates: First submitted 2018-06-30; First posted 2018-07-12 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Hemorrhage; Uterine Atony
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia | interventions — Carboprost; Methylergonovine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 15-methyl prostaglandin F2α (Active Comparator): IM Carboprost followed by Methylergonovine if needed.
  Interventions: Drug: 15-methyl prostaglandin F2α; Drug: Methylergonovine Maleate
- Methylergonovine Maleate (Active Comparator): IM Methylergonovine followed by Carboprost if needed.
  Interventions: Drug: 15-methyl prostaglandin F2α; Drug: Methylergonovine Maleate

INTERVENTIONS:
Drug: 15-methyl prostaglandin F2α — Participants will receive standard intraoperative care including an infusion of oxytocin immediately postpartum. If a second-line uterotonic is requested, patients randomized to the "carboprost" study group will receive an intramuscular dose of 0.25mg (1mL) carboprost. If another second-line uterotonic is requested, the patients will receive 0.2mg (1mL) intramuscular methylergonovine.
  Other Names: Carboprost
Drug: Methylergonovine Maleate — Participants will receive standard intraoperative care including an infusion of oxytocin immediately postpartum. If a second-line uterotonic is requested, patients randomized to the "methergine" study group will receive an intramuscular dose of 0.2mg (1mL) methylergonovine. If another second-line uterotonic is requested, the patients will receive 0.25mg (1mL) intramuscular carboprost.
  Other Names: Methylergonovine

SUMMARY:
The aim of this study is to evaluate in a randomized fashion the comparative efficacy of two second-line medications, methylergonovine and carboprost for treating atonic postpartum hemorrhage (PPH). The investigators hypothesize that administration of methylergonovine will produce superior uterine tone to carboprost in atonic PPH.

DETAILED DESCRIPTION:
Primary postpartum hemorrhage (PPH) is defined by the American College of Obstetricians and Gynecologists as a cumulative blood loss of >1000 mL within 24 hours of the birth process. PPH remains a leading source of maternal morbidity and mortality worldwide with uterine atony identified as the underlying cause in up to 80% of cases. Between 1994 and 2006, the rate of PPH increased by 26% in the United States, raising further concern for this problem.

Treatment of PPH typically begins with administration of exogenous oxytocin, a hormone responsible for uterine contraction. When postpartum bleeding persists despite oxytocin administration, a multidisciplinary approach combining mechanical, pharmacologic, and surgical measures is indicated. Approximately 3-25% of PPH cases require a second-line uterotonic agent in addition to oxytocin, with the two most commonly administered second-line agents in the U.S.A. being methylergonovine maleate (methylergonovine) and 15-methyl prostaglandin F2α (carboprost). The comparative efficacy of these two drugs is unknown and the most recent American College of Obstetricians and Gynecologists Practice Bulletin makes no recommendation on which second-line uterotonic agents to administer preferentially in the absence of contraindications.

This study will evaluate in a randomized fashion the comparative efficacy of methylergonovine and carboprost for treating atonic PPH. Patients undergoing non-emergent cesarean section (C/S) with uterine atony and no contraindications to either drug will be randomized to receive one of the two equivalent agents in a blinded fashion after oxytocin. After ten minutes, their uterine tone will be assessed by the obstetrician and reported on a 0-10 point scale.

A power calculation was performed to detect a mean difference in uterine tone between groups of 1 point on a 0-10 point scale with 80% power and significance level of 0.05. The investigators estimate 37 patients will be required in each arm. Allowing for a 20% rate of withdrawals or missing information, a total of 100 patients will be enrolled in this study.

Investigators will adhere to the FDA Expedited Safety Requirements in reporting any adverse event that is serious, unexpected, and associated with the use of the study drugs. Any such adverse event will be reported to the study site Institutional Review Board (IRB) and serious events will prompt the study to be halted until further discussion with the IRB.

ELIGIBILITY:
Inclusion Criteria:

* non-emergent cesarean delivery
* ASA I-III
* postpartum hemorrhage deemed the result of uterine atony (uterine atony at the time of delivery, despite the administration of oxytocin)

Exclusion Criteria:

* non-English speaking patients requiring an interpreter for urgent, unscheduled delivery
* any hypertensive disorder
* cardiovascular disease
* asthma
* refusal of transfused blood products
* coagulopathy or abnormal coagulation lab values
* hypersensitivity to methylergonovine maleate or 15-methyl prostaglandin
* known or suspected delayed postpartum hemorrhage after leaving the operating room

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naida M Cole, MD, Principal Investigator — Brigham and Women's Hospital, 75 Francis Street, Boston MA 02115
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data from this study will be de-identified and prepared in an anonymous data pack to minimize the possibility of re-identification. In the interests of the public good, ethical transparency, and economic and scientific support of future research, the data pack will be available to all appropriate requestors. The data will be shared in a secure fashion to protect the privacy of participants.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available upon publication of the study and for 10 years thereafter.
Access Criteria: Data requestors will be required to provide a detailed IRB-approved study protocol, data collection tools to be used and planned statistical analysis to the data generator. Citation of the data generator will be required if the data is used in a peer-reviewed publication.

REFERENCES:
- [Derived] Cole NM, Kim JJ, Lumbreras-Marquez MI, Fields KG, Mendez-Pino L, Farber MK, Carusi DA, Toledo P, Bateman BT. Second-Line Uterotonics for Uterine Atony: A Randomized Controlled Trial. Obstet Gynecol. 2024 Dec 1;144(6):832-841. doi: 10.1097/AOG.0000000000005744. Epub 2024 Sep 26. PMID 39326051
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2019- April 2022
Period: Overall Study
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Started | 50 | 50
Completed | 49 | 48
Not Completed | 1 | 2
Not completed — Primary outcome not measured | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (5.6) | 34.4 (4.4) | 33.6 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 25 | 26 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 100

OUTCOME MEASURES:

1. Primary Outcome: Uterine Tone Score
Description: Uterine contractile tone will be measured on a 0-10 score as assessed by the obstetrician; 0 is 'no tone', 10 is 'perfect tone' or 'excellent tone'.
Time Frame: at 10 minutes following administration of the first study drug
Population: In the carboprost group, 50 participants were enrolled and data for 49 participants were analyzed since the primary outcome was not measured in 1 participant. In the methylergonovine group, 50 participants were enrolled and data for 48 were analyzed since 2 participants did not have the primary outcome measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Number analyzed (Participants) | 49 | 48
score on a scale | 4.7 (1.9) | 4.4 (1.8)

2. Secondary Outcome: Uterine Tone Score
Description: as for outcome 1
Time Frame: at 5 minutes following administration of the first study drug
Population: 50 participants were enrolled in the 15-methyl prostaglandin F2alpha group, and this secondary outcome was measured in all participants. 50 participants were enrolled in the methylergonovine group, but 1 did not have this secondary outcome (uterine tone score 5 minutes after administration of the first study drug) measured, therefore 49 were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Number analyzed (Participants) | 50 | 49
score on a scale | 6.8 (1.9) | 6.4 (1.9)

3. Secondary Outcome: Number of Subjects Receiving Additional Uterotonic
Description: An additional second-line uterotonic which is given in the operating room after administration of the first study drug
Time Frame: from time of delivery until surgery completion, approximately 1-2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Number analyzed (Participants) | 50 | 50
Participants | 17 | 15

4. Secondary Outcome: Number of Subjects Requiring Transfusion
Description: The need for RBC transfusion due to postpartum blood loss.
Time Frame: within the first 24 hours after delivery of the fetus
Measure: Count of Participants; unit: Participants
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Number analyzed (Participants) | 50 | 50
Participants | 2 | 3

5. Secondary Outcome: Number of Subjects Requiring Additional Intervention
Description: The need for an additional surgical or radiologic intervention to control postpartum hemorrhage
Time Frame: within the first 24 hours after delivery of the fetus
Measure: Count of Participants; unit: Participants
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Number analyzed (Participants) | 50 | 50
Participants | 4 | 5

6. Secondary Outcome: Quantitative Blood Loss (QBL)
Description: The total volume of blood loss (in mL), calculated as a conversion from the measured blood loss in weight into its equivalent volume. Weight of blood loss is measured on a QBL scale that weighs surgical drapes, towels, sponges and suction fluid.
Time Frame: from entry to exit from the OR, approximately 2 to 3 hours
Measure: Geometric Mean (95% Confidence Interval); unit: milliliters (mL)
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Number analyzed (Participants) | 50 | 50
milliliters (mL) | 713 [621 to 820] | 758 [636 to 903]

7. Secondary Outcome: Hematocrit Drop
Description: Comparison of the preoperative and first postoperative hematocrit values
Time Frame: from time of preoperative hematocrit value before delivery until time of first postoperative hematocrit (within 24 hours postoperatively).
Measure: Mean (Standard Deviation); unit: percentage of initial Hct
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Number analyzed (Participants) | 50 | 50
percentage of initial Hct | 28.3 (3.7) | 27.7 (5)

8. Secondary Outcome: Length of Hospital Stay
Description: Total duration of hospital stay (in days)
Time Frame: from day of surgery to day of hospital discharge, approximately 3 days in most cases
Measure: Geometric Mean (95% Confidence Interval); unit: days
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Number analyzed (Participants) | 50 | 50
days | 4.1 [3.7 to 4.6] | 4.4 [4.1 to 4.7]

9. Secondary Outcome: Number of Subjects Experiencing Severe Maternal Morbidity
Description: Any unplanned adverse reaction or event with clinical consequences (e.g., cardiovascular event, intubation, ICU admission, hypovolemic shock, transfusion reaction, or adverse study drug reaction)
Time Frame: from time of delivery until time of hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant from the time of delivery until 1 month postpartum.
Arm/Group | 15-methyl Prostaglandin F2α | Methylergonovine Maleate
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 14/50 | 13/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15-methyl Prostaglandin F2α (N=50) | Methylergonovine Maleate (N=50)
nausea (Gastrointestinal disorders) | 14 (14) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT03584854/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT03584854/SAP_003.pdf